CLINICAL TRIAL: NCT06985238
Title: A Pilot Study to Determine Safety and Feasibility of the Stratagen Quantitative Prostate MRI Platform as an Adjunct to Standard of Care MRI When Evaluating for Clinically Significant Prostate Cancer
Brief Title: Stratagen Quantitative Prostate MRI Platform Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stratagen Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ST-25-001
Record Dates: First submitted 2025-04-22; First posted 2025-05-22 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Stratagen Quantitative Prostate MRI Platform (Experimental)
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Will receive up to 15 minutes of additional MRI scan time during the existing prostate MRI imaging session.

SUMMARY:
The goal of this clinical trial is to assess the safety and feasibility of the Stratagen Quantitative Prostate MRI Platform when used in addition to the standard scans conducted during the existing prostate MRI sessions.

* What severe problems, if any, occur because of the use of the Stratagen Quantitative Prostate MRI Platform?
* Can the data collected be used to measure quantitative MRI parameters?

Participants will:

- Receive up to 15 minutes of additional MRI scan time during the existing prostate MRI imaging session.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a prostate that would be considered for biopsy
* Age 40-90 years
* PSA ≥ 2.5
* Subject has been informed of the nature of the study and has provided written informed consent

Exclusion Criteria:

* Contraindication for MRI
* Prostate biopsy within the previous 12 weeks
* Implant in the pelvis that may cause artifact on MRI (e.g. hip replacement)
* History of prostatectomy or other local prostate cancer therapy (e.g., cryotherapy or brachytherapy), or previous pelvic irradiation
* Currently enrolled in another investigational drug or device study that clinically interferes with this study
* Unable to comply with the study requirements or follow up schedule
* Any condition the Investigator believes would interfere with the intent of this study or would make participation not in the best interest of the subject

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety: no SAEs attributable to the Stratagen Quantitative Prostate MRI Platform, as determined by participating Investigator according to CTCAE guidelines | Beginning of MRI Scan to end of MRI scan (MRI Scan Visit, Day 0)
  All serious adverse events attributable to the Stratagen Quantitative Prostate MRI Platform will be reported.
• Feasibility: collection of the data necessary to produce measurable quantitative T1 and T2 relaxation times (milliseconds) maps (images) for at least 80% of pixels fully contained within the prostate for at least 80% of subjects | Beginning of MRI Scan to end of MRI scan (MRI Scan Visit, Day 0)

CONTACTS AND LOCATIONS:
Locations (1):
- Urology Clinic at Sawgrass, Rochester, New York, United States